CLINICAL TRIAL: NCT07187505
Title: Venetoclax Plus All-Trans Retinoic Acid and Arsenic Trioxide in Newly Diagnosed Acute Promyelocytic Leukemia With Hyperleukocytosis: A Prospective Single-Arm Study
Brief Title: Venetoclax Combined With ATRA and ATO in Hyperleukocytic Acute Promyelocytic Leukemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Zhangbiao Long, Principal Investigator, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJ 2025-03-57(1)
Record Dates: First submitted 2025-09-06; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Promyelocytic Leukemia (APL)
Keywords: Venetoclax; All-Trans Retinoic Acid (ATRA); Arsenic Trioxide (ATO); Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — venetoclax; Tretinoin; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm: Venetoclax + ATRA + ATO (Experimental): Patients in this arm will receive a combination regimen consisting of venetoclax, all-trans retinoic acid (ATRA), and arsenic trioxide (ATO) as induction therapy, followed by consolidation according to protocol. The regimen is designed for newly diagnosed acute promyelocytic leukemia (APL) with hyperleukocytosis.
  Interventions: Drug: Venetoclax; Drug: All-trans retinoic acid; Drug: Arsenic Trioxide (ATO)

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is a selective BCL-2 inhibitor administered orally once daily. The dose will be adjusted according to the study protocol and patient tolerance.
  Other Names: Venclexta
Drug: All-trans retinoic acid — All-Trans Retinoic Acid (ATRA) is administered orally, twice daily, as part of standard induction and consolidation therapy for acute promyelocytic leukemia.
  Other Names: Tretinoin; Vesanoid
Drug: Arsenic Trioxide (ATO) — Arsenic Trioxide (ATO) is administered intravenously once daily, in combination with ATRA and venetoclax, during induction and consolidation therapy.
  Other Names: Trisenox

SUMMARY:
This study aims to evaluate the safety and effectiveness of combining venetoclax with all-trans retinoic acid (ATRA) and arsenic trioxide (ATO) in patients with newly diagnosed acute promyelocytic leukemia (APL) who have very high white blood cell counts. APL is a rare type of blood cancer, and patients with high white blood cell levels often face serious complications. Current treatments with ATRA and ATO are effective, but the outcomes for patients with high white blood cells remain poor. This study will test whether adding venetoclax, a drug that helps leukemia cells die, can improve treatment results.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE 1. To evaluate the efficacy of the venetoclax + ATRA + ATO regimen, as defined by complete remission (CR), complete remission with incomplete hematologic recovery (CRi), and morphological leukemia-free state (MLFS).

________________________________________ SECONDARY OBJECTIVES

1. To evaluate long-term effectiveness and durability of the regimen, as defined by 1-year overall survival (OS), 1-year event-free survival (EFS), and overall response rate (ORR).
2. To evaluate the safety of the regimen, as defined by Grade 3-4 clinical adverse events (AEs), incidence of laboratory abnormalities, differentiation syndrome, and treatment-related mortality (TRM).
3. To assess transfusion requirements (red blood cells and platelets) during induction.

   ________________________________________ OUTLINE
   * Newly diagnosed hyperleukocytosis group: Patients with baseline WBC >10 × 10⁹/L will receive venetoclax + ATRA + ATO as induction therapy.
   * Secondary hyperleukocytosis group: Patients who develop WBC >10 × 10⁹/L for ≥3 consecutive days during therapy will receive venetoclax added dynamically to ATRA + ATO.

   Induction regimen:
   * Venetoclax (VEN): 100 mg orally once daily on days 1-7. For patients with WBC >100 × 10⁹/L, administer 50 mg on days 1-2, then escalate to 100 mg on days 3-7.
   * All-Trans Retinoic Acid (ATRA): 25 mg/m² orally per day (divided doses), on days 1-28.
   * Arsenic Trioxide (ATO): 0.15 mg/kg intravenously once daily, on days 1-28.

   Assessment:
   * Complete blood counts monitored regularly.
   * Bone marrow evaluation on days 14 and 28.
   * One treatment cycle lasts 28 days.

   Response evaluation:
   * On day 21 of the first cycle, bone marrow assessment will be performed.
   * If CR, CRi, or MLFS is not achieved, induction with the same regimen will continue for one additional cycle.
   * Patients failing to achieve remission after two cycles will be withdrawn from the study.
   * Patients achieving remission will proceed to consolidation and maintenance therapy according to investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute promyelocytic leukemia (APL) according to bone marrow morphology and immunophenotyping, consistent with the WHO 2016 diagnostic criteria.
2. Age ≥14 years, both male and female patients are eligible.
3. Adequate organ function, defined as:

   3.1 Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3 × upper limit of normal (ULN);

   3.2 Total serum bilirubin ≤1.5 × ULN;

   3.3 Creatinine clearance ≥30 mL/min;

   3.4 Serum cardiac enzymes <2.0 × ULN.
4. Signed informed consent obtained from the patient or a legally authorized representative.
5. White blood cell (WBC) count >10 × 10⁹/L at initial diagnosis, or WBC >10 × 10⁹/L during treatment.

Exclusion Criteria:

1. Diagnosis of acute non-promyelocytic leukemia, myeloid sarcoma, or chronic myeloid leukemia in accelerated or blast phase.
2. Known hypersensitivity to any drug included in the study regimen.
3. Pregnant or breastfeeding women, and women of childbearing potential who are unwilling to use effective contraception during the study treatment period.
4. Presence of organic heart disease, such as uncontrolled or symptomatic arrhythmia, congestive heart failure, or myocardial infarction within 6 months prior to screening that resulted in clinical symptoms or impaired cardiac function (NYHA class ≥III).
5. Concurrent malignancies, except for:

   5.1 Malignancies treated with curative intent (e.g., hematopoietic stem cell transplantation) and with no known active disease for ≥5 years before enrollment;

   5.2 Adequately treated non-melanoma skin cancer or malignant lentigo without evidence of disease, even if diagnosed <3 years before enrollment;

   5.3 Adequately treated carcinoma in situ without evidence of disease, even if diagnosed <3 years before enrollment.
6. Patients with acquired immunodeficiency syndrome (AIDS) or syphilis, or those with active hepatitis B (detectable HBV DNA) or active hepatitis C infection.
7. Any concurrent medical condition or disease that may interfere with study procedures or outcomes, or that may pose an unacceptable risk to the participant as determined by the investigator (e.g., active systemic infection).
8. Inability to understand or comply with the study protocol.
9. Participation in another clinical study within 1 month prior to enrollment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Early Mortality (Day 0-30) | 30 days
  Proportion of patients who die from any cause within 30 days after treatment initiation.

SECONDARY OUTCOMES:
Incidence of Complications | 30 days
  Proportion of patients experiencing severe complications related to induction therapy.
Event-Free Survival (EFS) | Up to 2 years
  Time from enrollment to treatment failure, relapse, or death from any cause.
Overall Response Rate (ORR) | At 3 months after induction therapy
  Proportion of patients achieving overall response, defined as complete remission (CR) plus partial remission (PR).

OTHER OUTCOMES:
Changes in Daily White Blood Cell Count During Induction | 30 days
  Monitoring daily white blood cell (WBC) counts during the induction phase.
Incidence of Laboratory Abnormalities | From enrollment through 2 years.
  Frequency of grade 3-4 abnormal laboratory test results according to CTCAE.
Incidence of Differentiation Syndrome | 30 days
  Proportion of patients developing differentiation syndrome during induction therapy.
Frequency of Blood Product Transfusion | 30 days
  Number of blood or platelet transfusions during induction therapy.
Volume of Blood Product Transfusion | 30 days
  Total amount of blood or platelet transfused (units or mL) during induction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhangbiao Long, Study Chair — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- Department of Hematology, The First Affiliated Hospital of Anhui Medical University, 218 Jixi Road, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including demographic information, baseline characteristics, efficacy outcomes, and safety data, will be shared. Data will be provided to qualified researchers for the purpose of academic research. Access will require submission of a research proposal and approval by the study steering committee, as well as signing a data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting documents will be available beginning 6 months after publication of the primary results and will remain available for 3 years.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the de-identified IPD and supporting documents. Requests should be submitted to the Principal Investigator by email. Proposals will be reviewed by the study steering committee, and access will be granted after approval and signing of a data access agreement.